CLINICAL TRIAL: NCT03318705
Title: Testing Latest Version of NidekRS3000Adv
Status: Completed | Type: Observational
Sponsor: Doheny Image Reading Center (Other)
Responsible Party: Principal Investigator, Kenneth Marion, Program Manager - Research, Doheny Image Reading Center
Other Study IDs: NIDEKRS3000ADV
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Device: RS3000Adv — Nidek RS3000Adv device to be used to take images which will allow measurement of vascularization in participants

SUMMARY:
The investigators would like to know if different imaging devices can improve the quality of images and visualization of imaged tissues. Also, the investigators would like to find out whether these changes are useful in the diagnosis and treatment of eye diseases. Using images of previous participants will allow us to demonstrate the advancement of different technologies, as well be used to allow comparisons between current technologies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* 18 years old or older

Exclusion Criteria:

* Those suffering from head, neck or other injury which makes them unable to position themselves in head restraint for imaging
* subjects who are unable to maintain retinal fixation on a specified target
* subjects unable to achieve sufficient pupil dilation and alignment stability for imaging to take place
* subjects with media opacity which preclude high quality imaging will be excluded.
* vulnerable subjects
* subjects under 18
* pregnant subjects
* economically and educationally disadvantaged subjects
* decision impaired subjects
* homeless subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Control subjects with no ocular problems, with whom no record review will be conducted, but imaging will be conducted with study devices.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Ocular vascularization | 1 year
  Nidek RS3000Adv device to be used to take images which will allow measurement of vascularization in participants

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Sadda, MD, Principal Investigator — Doheny Eye Institute
Locations (1):
- Doheny Eye Centers UCLA, Pasadena, California, United States